CLINICAL TRIAL: NCT04524143
Title: The Acute Effect of Cervical Mobilization on Balance and Gait in Patients With Idiopathic Parkinson's Disease
Brief Title: The Acute Effect of Cervical Mobilization in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ayla fil balkan, Assoc. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-180099
Record Dates: First submitted 2020-08-18; First posted 2020-08-24 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Cervical Spine; Postural Balance; Gait; Manual Therapies
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Other): There was no intervention in the control group during the study (At the end of study all patients were received home-based exercise)
  Interventions: Other: control
- mobilization group (Experimental): Cervical mobilization was applied to the mobilization group. Cervical mobilization techniques were applied for 10 minutes in the supine position. (At the end of study all patients were received home- based exercise)
  Interventions: Other: cervical mobilization; Other: control

INTERVENTIONS:
Other: cervical mobilization — Cervical mobilization techniques were applied in the study. Within the scope of application; rotation with traction, lateral gliding, anterior-posterior gliding with traction, bridging and stroking techniques to the paravertebral muscles were used. Mobilization were performed at grade A (mobilization in painless joint range) and grade B (continuous stretching at the end of the joint range). The mobilization were applied during 10 minutes.
  At the end of study all patients were received home-based exercise tailored to each individual's needs which include stretching, strengthening, balance and gait exercise and posture exercise
  Arms: mobilization group
Other: control — There was no intervention in the control group during study. At the end of study all patients were received home-based exercise tailored to each individual's needs which include stretching, strengthening, balance and gait exercise and posture exercise

SUMMARY:
Patients with Idiopathic Parkinson's disease have balance and gait problems due to sensory and motor impairments. In the literature, there are lots of studies including various approaches for rehabilitation of these parameters such as sensory interventions, conservative treatments, neurophysiological approaches and motor imagery. However, taking into account of literature, there is no study investigating the effects on balance and gait of cervical mobilization by stimulating proprioceptors and vestibular receptors. Therefore, the aim of this study is to investigate the acute effect of cervical mobilization on balance and gait in patients with idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
Patients with Idiopathic Parkinson's disease have balance and gait problems due to sensory and motor impairments. In the literature, there are lots of studies including various approaches for rehabilitation of these parameters such as sensory interventions, conservative treatments, neurophysiological approaches and motor imagery. The posture of the cervical region is impaired by the findings of the disease such as rigidity, flexor posture and loss of axial rotation. Considering that the cervical region is rich in proprioceptors and one of the key points for the vestibular system, interventions to this area can be thought to contribute to postural control and gait. However, taking into account of literature, there is no study investigating the effects on balance and gait of cervical mobilization by stimulating proprioceptors and vestibular receptors. Therefore, the aim of this study is to investigate the acute effect of cervical mobilization on balance and gait in patients with idiopathic Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Idiopathic Parkinson's disease
* Being between the ages of 50-80
* Patients scoring >24 on Standardized Mini Mental State Examination
* Modified Hoehn and Yahr stage 2-3
* No medication or dose changes during treatment
* Not participating in the physiotherapy and rehabilitation program in the last 6 months
* Volunteering to participate in the study

Exclusion Criteria:

* Vertebrobasilar insufficiency
* Other neurological diseases
* Postural hypotension, visual problems (which can not be compensated with the correct lens) or vestibular disorders that may affect balance
* Cardiopulmonary diseases that may affect gait
* Orthopedic problems (such as fracture, osteomyelitis, severe osteoporosis), advanced inflammatory arthritis, knee prothesis
* Uncontrolled dyskinesia or motor fluctuation
* Excessive use of alcohol or substance abuse
* Anticoagulant therapy, blood clotting diseases
* Long-term use of corticosteroids

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Static Posturography Assesment (NeuroCom® Balance Master® Systems) | Baseline and immediately after cervical mobilization
  Posturography measures postural stability statically and dynamically. Device has lots of test parameters such as Modified Clinical Test of Sensory Integration on Balance Test, limits of stability, rhythmic weight shift, weight bearing squat, unilateral stance, sit to stand, walk across, tandem walk, step/quick turn, step up/over and forward lunge. In addition to assesment, exercise training can also be given by posturography.
Dynamic Gait Index | Baseline and immediately after cervical mobilization
  It is a measurement tool that can be used to assess dynamic balance, gait, and risk for falls. Balance and walking pattern changes are scored during tasks such as changing gait speed, gait with vertical and horizontal head turns, pivot turn, step over obstacle, step around obstacles and climbing stairs.
  A four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function.Total score is 24 for this scale.

SECONDARY OUTCOMES:
Clinical Test of Sensory Integration on Balance | Baseline and immediately after cervical mobilization
  In this clinical test, which evaluates the static balance in the standing posture, there are 6 different parameters that are formed by a combination of three visual (eyes open, eyes closed and DOME) and two support surfaces (firm and foam floor). Oscillations are observed during the evaluation and it is expected to maintain each test position for 30 seconds
Functional Reach Test | Baseline and immediately after cervical mobilization
  It is used to evaluate dynamic equilibrium and anteroposterior stability. Test is performed with the participant in standing. It is the measure of the difference between arm's length with arms at 90° flexion and maximal forward reach. A score between 6-10 inches indicates a moderate risk for falls.
Tandem Stance Balance Test | Baseline and immediately after cervical mobilization
  In the tandem position, a person places one foot in front of the other and tries to maintain its balance in this position. The stance time is recorded.

OTHER OUTCOMES:
Mini-Mental State Examination | Baseline
  The Mini-Mental Status Examination offers a quick and simple way to quantify cognitive function and screen for cognitive loss.It tests the individual's orientation, attention, calculation, recall, language and motor skills. Each section of the test involves a related series of questions or commands. The individual receives one point for each correct answer. To give the examination, seat the individual in a quiet, well-lit room. Ask him/her to listen carefully and to answer each question as accurately as he/she can. Don't time the test but score it right away. To score, add the number of correct responses. The individual can receive a maximum score of 30 points. A score below 20 usually indicates cognitive impairment.
The Modified Hoehn and Yahr Scale | Baseline
  It is used to describe the symptom progression of Parkinson disease. It was designed to be a descriptive staging scale to evaluate both disability and impairment related to clinical disease progression. It was originally published in 1967 and included stages 1 through 5. Since then, a modified Hoehn and Yahr scale was proposed with the addition of stages 1.5 and 2.5 to help describe the intermediate course of the disease.
  Modified Hoehn and Yahr Staging
  STAGE 0 = No signs of disease. STAGE 1 = Unilateral disease. STAGE 1.5 = Unilateral plus axial involvement. STAGE 2 = Bilateral disease, without impairment of balance. STAGE 2.5 = Mild bilateral disease, with recovery on pull test. STAGE 3 = Mild to moderate bilateral disease; some postural instability; physically independent.
  STAGE 4 = Severe disability; still able to walk or stand unassisted. STAGE 5 = Wheelchair bound or bedridden unless aided.
Unified Parkinson's Disease Rating Scale | Baseline
  It is used to evaluate the symptoms of the disease and complications related to treatment. In this scale consisting of 4 parts, the scoring of each item is between 0-4 points. (I = Mental state, behavior and mental state, II = Activities of daily living, III = Motor examination, IV = Treatment complications). Parts I to III are scored on a 0-4 rating scale. Part IV is scored with yes and no ratings. Higher scores indicate increased severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Özcan, MSc, Principal Investigator — Çankırı Karatekin University; Gül Yalçın Çakmaklı, Assoc. Prof, Study Director — Hacettepe University; Ayla Fil Balkan, Assoc. Prof, Study Chair — Hacettepe University; Bülent Elibol, Prof. Dr., Study Chair — Hacettepe University; Songül Aksoy, Prof. Dr., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noll DR. Management of falls and balance disorders in the elderly. J Am Osteopath Assoc. 2013 Jan;113(1):17-22. PMID 23329802
- [Background] Lopez D, King HH, Knebl JA, Kosmopoulos V, Collins D, Patterson RM. Effects of comprehensive osteopathic manipulative treatment on balance in elderly patients: a pilot study. J Am Osteopath Assoc. 2011 Jun;111(6):382-8. doi: 10.7556/jaoa.2011.111.6.382. PMID 21771924
- [Background] Wells MR, Giantinoto S, D'Agate D, Areman RD, Fazzini EA, Dowling D, Bosak A. Standard osteopathic manipulative treatment acutely improves gait performance in patients with Parkinson's disease. J Am Osteopath Assoc. 1999 Feb;99(2):92-8. doi: 10.7556/jaoa.1999.99.2.92. PMID 10079641
- [Background] Brink EE, Jinnai K, Hirai N, Wilson VJ. Cervical input to vestibulocollic neurons. Brain Res. 1981 Jul 27;217(1):13-21. doi: 10.1016/0006-8993(81)90181-5. PMID 6266589
- [Background] Mergner T, Siebold C, Schweigart G, Becker W. Human perception of horizontal trunk and head rotation in space during vestibular and neck stimulation. Exp Brain Res. 1991;85(2):389-404. doi: 10.1007/BF00229416. PMID 1893987
- [Background] Haavik-Taylor H, Murphy B. Cervical spine manipulation alters sensorimotor integration: a somatosensory evoked potential study. Clin Neurophysiol. 2007 Feb;118(2):391-402. doi: 10.1016/j.clinph.2006.09.014. Epub 2006 Nov 29. PMID 17137836
- [Background] Haavik H, Murphy B. The role of spinal manipulation in addressing disordered sensorimotor integration and altered motor control. J Electromyogr Kinesiol. 2012 Oct;22(5):768-76. doi: 10.1016/j.jelekin.2012.02.012. Epub 2012 Apr 6. PMID 22483612
- [Background] Holt KR, Haavik H, Elley CR. The effects of manual therapy on balance and falls: a systematic review. J Manipulative Physiol Ther. 2012 Mar-Apr;35(3):227-34. doi: 10.1016/j.jmpt.2012.01.007. Epub 2012 Feb 17. PMID 22343006